CLINICAL TRIAL: NCT03667092
Title: Pilot Study for Measuring Molecular Biomarkers and Their Capacity to Characterize Radionuclide Therapy With Lu-177 DOTATATE) in Metastatic G1-G2 Neuroendocrine Midgut Tumors
Brief Title: Exploration of Molecular Biomarkers for Lu-177 DOTATATE Therapy in Midgut Neuroendocrine Tumor
Acronym: GENEBIOLuNET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC31/17/0356
Record Dates: First submitted 2018-07-27; First posted 2018-09-12 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Midgut Neuroendocrine Tumors
Keywords: Lu-177 Dotatate; transcript analysis and variation; molecular biomarkers; midgut neuroendocrine tumors
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Non-drug intervention type (Experimental): Exploration of gene transcript variation on seriate blood samples before treatment, before and after the 2nd and the 4th Lu-Dotatate injection and before and after the 6 month post treatment follow-up.
  Measures of stability and reproducibility of selected gene transcripts and miRNA as radio sensitivity genes or progressive metastatic midgut neuroendocrine tumors genetic signatures before and during Lu-177 Dotatate internal vectorized therapy, as well as on the 6-month follow-up.
  Interventions: Biological: non-drug intervention type

INTERVENTIONS:
Biological: non-drug intervention type — 8 peripheral blood samples (8x5ml) will be obtained at different times ; before, during and after treatment
  Other Names: Blood samples

SUMMARY:
Midgut neuroendocrine tumours present an increasing incidence and poor survival at 5 years with limited therapeutic options for metastatic, non-operable cases. Lu-177 Dotatate, targeting somatostatin receptors, is an internal vectorized radiotherapy using Lu-177, an ideal radionuclide for peptide radionuclide therapy. In NETTER-1 phase III randomized clinical trial, Lu-177 Dotatate proved its superiority in increasing progression free survival for midgut neuroendocrine tumors. This study hypothesize that finding biomarkers of individual radio sensitivity for this type of internal vectorized therapy would allow treatment personalization. The protocol aim at studying transcript variations induced by this therapy.

DETAILED DESCRIPTION:
Internal vectorized therapy using Lu-177 Dotatate (abbreviated peptide receptor radionuclide therapy) was recently shown to improve progression free survival and response in metastatic progressive midgut neuroendocrine tumors (NETTER-1 phase III trial).

Lu-177 Dotatate is administered as a series of four consecutive intra veinous injections of an activity of 7.4 gigabequerel every 8 weeks.

In order to identify potential biomarkers of radio sensitivity to Lu-177 Dotatate, investigators aim to study the stability of gene/miRNA transcripts in the absence of Lu-177 Dotatate or at 6 months after treatment as well as the variations in transcript analysis after 2 Lu-177 Dotatate injections and at the end of the treatment.

Transcript variation analysis will be confronted and correlated with peripheral blood pharmacokinetic studies aimed at calculating time activity curves and provide biodosimetry information; other correlations with imaging modalities assessment of dosimetry or disease response to treatment or toxicity effects induced by Lu-177 Dotatate will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years old; histopathologically confirmed grade 1-2 midgut neuroendocrine tumor with documented progression during the year preceding inclusion upon RECIST criteria on computerized tomography, Octreoscan or Ga-68 positron emission tomography/computerized tomography
* Patients having an indication for Lu-177 Dotatate treatment validated during multidisciplinary meeting coordinated by Pr Rosine Guimbaud under RENATEN coordination;
* Measurable target lesions upon RECIST criteria
* Patients on somatostatin analogues treatment. Every somatostatin analogue injection should be organized to be administered 24 to 48 hours after each injection of Lu-177 Dotatate.
* All patients should be in a clinical state allowing them to continue treatment.
* Social security affiliation is mandatory.

Exclusion Criteria:

* Patients on chemotherapy or other targeted therapy within the 4 months preceding peptide receptor radionuclide therapy
* Fertile patients refusing active contraception ; pregnancy.
* Patients with prior chemotherapy or peptide receptor radionuclide therapy administration
* Patients with uncontrollable psychotic disorders
* Renal hepatic and medullary insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2024-05-22 (Actual); Study Completion 2024-05-22 (Actual)

PRIMARY OUTCOMES:
Peptide receptor radionuclide therapy radio-induction variation of radiosensibility/reparation genes | Change from before at during treatment
  Variations in gene transcripts will be registered and processed by a bio-informatician

SECONDARY OUTCOMES:
Evaluation of gene transcript variations | during treatment and until 48 hours after treatment
  Analysis of gene transcript variation by quantitative real-time polymerase chain reaction
Evaluation of interindividual variability with NONMEN software | during treatment and until 48 hours after treatment
  Analysis of Lu-177 DOTATATE plasma concentration during treatment and 48 hours after treatment
Evaluation of therapeutic response according to RECIST criteria | 6 months post therapy
  Correlation between gene variations and the therapeutic response assessed on RECIST criteria

CONTACTS AND LOCATIONS:
Overall Officials: Lavinia VIJA, MD, PhD, Study Chair — University Hospital, Toulouse
Locations (1):
- CHU de Toulouse, Toulouse, France, France